CLINICAL TRIAL: NCT02996058
Title: Dexmedetomidine Sedation in Pediatric Intensive Care Unit
Brief Title: Safety And Efficacy Of Dexmedetomidine Sedation In Intubated Mechanically Ventilated Infants With Respiratory Failure
Acronym: DEXinPICU
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/00436
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEX I 0.35µg/kg /h (Active Comparator): the infants will receive a maintenance dose of 0.35µg/kg /h of Dexmedetomidne without a loading dose and guided by the assessed sedation scale
  Interventions: Drug: Dexmedetomidine 0.35µg/kg /h
- DEX II 0.5µg/kg /h (Active Comparator): the infants will receive a maintenance dose of 0.5µg/kg /h of Dexmedetomidne without a loading dose and guided by the assessed sedation scale.
  Interventions: Drug: Dexmedetomidine 0.5µg/kg /h

INTERVENTIONS:
Drug: Dexmedetomidine 0.35µg/kg /h — the infants will receive a maintenance dose of 0.35µg/kg /h of Dexmedetomidne without a loading dose and guided by the assessed sedation scale
  Other Names: Precedex
  Arms: DEX I 0.35µg/kg /h
Drug: Dexmedetomidine 0.5µg/kg /h — the infants will receive a maintenance dose of 0.5µg/kg /h of Dexmedetomidne without a loading dose and guided by the assessed sedation scale
  Other Names: Precedex
  Arms: DEX II 0.5µg/kg /h

SUMMARY:
Dexmedetomidine is a highly selective α2-agonist with hypnotic, analgesic, and anxiolytic properties. Despite off-label administration, dexmedetomidine has found a niche in critically ill mechanically ventilated neonates and infants because of its minimal effects on respiratory function at sedative doses, facilitating early extubation and fast-track postoperative care.

DETAILED DESCRIPTION:
Critically ill children require sedation for comfort and to facilitate mechanical ventilation and interventions. The ideal sedative agent for use in critically ill children has to be effective and short-acting, of rapid onset of action, lacks active metabolites, does not accumulate in patients with renal or hepatic dysfunction, has minimal to no cardiovascular or respiratory adverse effects, and has few drug interactions.

Dexmedetomidine is a highly selective α2-agonist with hypnotic, analgesic, and anxiolytic properties. Despite off-label administration, dexmedetomidine has found a niche in critically ill mechanically ventilated neonates and infants because of its minimal effects on respiratory function at sedative doses, facilitating early extubation and fast-track postoperative care.

The only FDA approved indication of dexmedetomidine is sedation of intubated mechanically ventilated adults for less than 24h. However, the literature is full of many research studies that investigated the use off-lable use of dexmedetomidine for sedation more than 24h in both adult and pediatric population and proved its safety and effectiveness.

The aim of this study will be to investigate the safety and efficacy of dexmedetomidine in two different doses in sedation for critically ill mechanically ventilated infants with respiratory failure for 72h duration.

ELIGIBILITY:
Inclusion Criteria:

* Infants (1-12 months).
* Respiratory failure/
* Requiring PICU admission and mechanical ventilation up to 72h.

Exclusion Criteria:

* Significant renal, hepatic, endocrine or metabolic disease.
* 2nd or 3rd degree heart block.
* hypotension or bradycardia (defined as any value outside the normal range from the patient's age).

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
University of Michigan sedation scale | 72H
  The university of Michigan sedation scale (UMSS) will be assessed every hour

SECONDARY OUTCOMES:
The blood pressure | 72h
  The invasive arterial blood pressure will be recorded every hour
The heart rate | 72h
  The heart rate will be recorded every hour.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in anesthesia and intensive care, faculty of medicine, Assiut university, Egypt
Locations (1):
- Pediatric hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No